CLINICAL TRIAL: NCT03490682
Title: Effect of Labour on the Gastric Emptying of a Light Meal
Brief Title: Gastric Emptying During the Labour
Acronym: VGObstetric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL17_0863; 2017-A03605-48 (Other: ID-RCB)
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy; Healthy Volunteers; Parturition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Non-pregnant control (Active Comparator): adult females aged less than 40 years, not currently pregnant, without significant medical history (American Society of Anesthesiologists ASA 1), fasting for at least 6 hours for solids and 1 hour for clear fluids.
  Interventions: Other: Ultrasound assessment of gastric emptying of a flavoured yoghourt.
- Pregnant control (Active Comparator): adult females aged less than 40 years, pregnant in the third trimester (gestation greater than 32 weeks on the day of the study) according to dates and the calculation of term established at the start of the pregnancy by an obstetrician, without significant medical history (American Society of Anesthesiologists ASA 1), fasting for at least 6 hours for solids and I hour for clear fluids.
  Interventions: Other: Ultrasound assessment of gastric emptying of a flavoured yoghourt.
- Analgesia (Experimental): adult females aged less than 40 years, without significant medical history (American Society of Anesthesiologists ASA 1), in labour in the delivery suite, with a working epidural, having consumed solid food more than 6 hours before inclusion in the study and clear fluids more than 1 hour before inclusion in the study, and allowed to ingest solids during labour (cervical dilatation strictly less than 8cm) conforming to local protocols.
  Interventions: Other: Ultrasound assessment of gastric emptying of a flavoured yoghourt.
- Parturient (Experimental): adult females aged less than 35 years, without significant medical history (American Society of Anesthesiologists ASA 1), in labour in the delivery suite, without any epidural analgesia, having consumed solid food more than 6 hours before inclusion in the study and clear fluids more than 1 hour before inclusion in the study, and allowed to ingest solids during labour (cervical dilatation strictly less than 8cm) conforming to local protocols.
  Interventions: Other: Ultrasound assessment of gastric emptying of a flavoured yoghourt.

INTERVENTIONS:
Other: Ultrasound assessment of gastric emptying of a flavoured yoghourt. — Each participant will be placed on a table, in the semi-recumbent position with elevation of the head at 45° and a first ultrasound examination will be performed. After that, the participant will be invited to eat a test meal (flavoured yoghurt) in 5 minutes. An ultrasound examination of the antrum allowing measurement of the antral area will be performed at 15, 60, 90 and 120 minutes after the end of the ingestion of the test meal. The participant must stay in the semi-recumbent position during the total duration of the study. The non-invasive ultrasound measurement, of the antral cross-sectional area is performed using a Sonosite ultrasound equiped with a 2 -5.5MHz probe. The diameters (longitudinal D1 and anteroposterior D2) of the antrum are measured in the sagittal plane passing by the abdominal aorta and the left lobe of the liver. The value of the antral cross-sectional area is given by the formula : Antral area = π x D1 x D2 / 4.

SUMMARY:
Current recommendations permit the ingestion of all clear fluids (water, apple juice, black coffee..) during labour. However, regarding food during labour, the recommendations vary. British and European guidelines permit the ingestion of low-residue food during labour whilst guidelines from the United States prohibit having any solid food during labour. The reason for this variation in recommendations is the lack of data on gastric emptying during labour with a conservative approach adopted due to the fear of delayed gastric emptying increasing the risk of regurgitation and pulmonary aspiration in the case of general anaesthesia. This study aims, therefore, to evaluate if the gastric emptying of a light meal is slowed down during labour, using a validated, non-invasive ultrasound method, in four groups of women : Women in labour with epidural analgesia (Analgesia group), women in labor without any epidural analgesia (Parturient group), women in the third trimester of pregnancy (Pregnant group) and women who are not currently pregnant (Non-pregnant control group). The investigator propose the hypothesis that the gastric emptying of a light, solid meal is slowed by 30% during labour under epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

Informed consent must have been signed. The last consumption of solids will have taken place more than 6 hours before the start of the study, the last consumption of clear fluids will have taken place more than 1 hour before the start of the study, in the three groups.

* Non-pregnant control group : adult females less than 40 years old with no significant medical history (American Society of Anesthesiologists ASA class 1)
* Pregnant group : adult females less than 40 years old with no significant medical history (American Society of Anesthesiologists ASA class 1) in the third trimester of pregnancy (gestation greater than 32 weeks on the day of the study).
* Analgesia group : adult females less than 40 years old with no significant medical history (American Society of Anesthesiologists ASA class 1, in labour in the delivery room, receiving effective epidural analgesia, having an empty stomach on the initial ultrasound examination, and authorised to ingest solid foods during labour (cervical dilatation strictly less than 8cm) according to local guidelines.
* Parturient group : adult females less than 35 years old with no significant medical history (American Society of Anesthesiologists ASA class 1, in labour in the delivery room, no epidural analgesia, having an empty stomach on the initial ultrasound examination, and authorised to ingest solid foods during labour (cervical dilatation strictly less than 8cm) according to local guidelines

Exclusion Criteria:

* Refusal to participate in this study
* Patient unable to speak French
* Oesophageal, duodenal or gastric medical or surgical history Pregnant group : Threatened premature labour, multiple pregnancy, pathological pregnancy

Analgesia and Parturient groups :

* gestation less than 38 weeks
* multiple pregnancy
* All pathology of the pregnancy or complication during labour
* Delivery
* Patient admission for therapeutic interruption of the pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
determination of the rate of gastric emptying of a light meal in the 3 groups of women | 15 min after the ingestion of a flavoured yoghurt
  The rate of gastric emptying will be calculated using the following formula : Rate = [(Antral area at 90 min / Antral area at 15 min)-1] x 100
determination of the rate of gastric emptying of a light meal in the 3 groups of women | 90 min after the ingestion of a flavoured yoghurt
  The rate of gastric emptying will be calculated using the following formula : Rate = [(Antral area at 90 min / Antral area at 15 min)-1] x 100

SECONDARY OUTCOMES:
Comparison of the rate of gastric emptying between the Control group and the Pregnancy group | 15 min after the ingestion of a flavoured yoghurt
  The rate of gastric emptying will be calculated using the following formula : Rate = [(Antral area at 90 min / Antral area at 15 min)-1] x 100
Comparison of the rate of gastric emptying between the Control group and the Pregnancy group | 90 min after the ingestion of a flavoured yoghurt
  The rate of gastric emptying will be calculated using the following formula : Rate = [(Antral area at 90 min / Antral area at 15 min)-1] x 100
Calculation of the sonographic rate of gastric emptying in the three groups of women. | 15 min after the ingestion of a flavoured yoghurt
  In each group, the rate of gastric emptying will be calculated using the following formula : Rate = [(Antral area at 60 min / Antral area at 15 min)-1] x 100
Calculation of the sonographic rate of gastric emptying in the three groups of women. | 60 min after the ingestion of a flavoured yoghurt
  In each group, the rate of gastric emptying will be calculated using the following formula : Rate = [(Antral area at 60 min / Antral area at 15 min)-1] x 100
The rate of women having an empty stomach after the ingestion of the test meal in each group. | 90 min
  Empty stomach will be defined by the lack of ultrasound visualization of any content in the semirecumbent position with antral area ≤ 505 mm² in groups Parturient and Pregnancy, and by the lack of visualization of any content with antral area ≤ 340 mm² in the Control group, 90 and 120 min after ingestion of the test meal.
The rate of women having an empty stomach after the ingestion of the test meal in each group. | 120 min
  Empty stomach will be defined by the lack of ultrasound visualization of any content in the semirecumbent position with antral area ≤ 505 mm² in groups Parturient and Pregnancy, and by the lack of visualization of any content with antral area ≤ 340 mm² in the Control group, 90 and 120 min after ingestion of the test meal.
Comparison of the rate of gastric emptying between the Analgesia group and the Parturient group | 15 min after the ingestion of a flavoured yoghurt
  The rate of gastric emptying will be calculated using the following formula : Rate = [(Antral area at 90 min / Antral area at 15 min)-1] x 100
Comparison of the rate of gastric emptying between the Analgesia group and the Parturient group | 90 min after the ingestion of a flavoured yoghurt
  The rate of gastric emptying will be calculated using the following formula : Rate = [(Antral area at 90 min / Antral area at 15 min)-1] x 100

CONTACTS AND LOCATIONS:
Overall Officials: Lionel BOUVET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

REFERENCES:
- [Background] Bouvet L, Schulz T, Piana F, Desgranges FP, Chassard D. Pregnancy and Labor Epidural Effects on Gastric Emptying: A Prospective Comparative Study. Anesthesiology. 2022 Apr 1;136(4):542-550. doi: 10.1097/ALN.0000000000004133. PMID 35103759